CLINICAL TRIAL: NCT04785404
Title: Primary Versus Secondary Closure of Stoma-Reversal Skin Wound: Randomized Controlled Trial
Brief Title: Primary Versus Secondary Closure of Stoma-Reversal Skin Wound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayub Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AyubTH
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Wound Infection
Keywords: skin closure; stoma reversal
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Intervention Model Description: patients will be randomly distributed to two groups. Group A patients will have skin wounds stithed after stoma reversal while in secondary closure group B, wound will be allowed to heal by secondary intention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- primary skin closure (Experimental): in this group, skin wound will be primarily closed
  Interventions: Procedure: primary skin closure
- secondary skin closure (No Intervention): skin will be left open to heal by secondary intention

INTERVENTIONS:
Procedure: primary skin closure — skin will be stitched after stoma reversal to heal by primary intention
  Arms: primary skin closure

SUMMARY:
to compare infection rate stoma reversal skin wound after primary or secondary closure

DETAILED DESCRIPTION:
There will be two groups. In group A, skin will be stitched with prolene while in group B skin will be left open to follow up till 1 month and wound observed for infection according to CDC guidelines.

ELIGIBILITY:
Inclusion Criteria:

* . All patients who undergo ileostomy or colostomy reversal will be included

Exclusion Criteria:

* included patients with reversal of stoma through laparatomy, post-operative anastomotic leak and co-morbidities like diabetes, Chronic liver disease, chronic kidney disease etc

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
surgical site infection | 30 days
  skin wound infection at surgical site will be observed on CDC guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Zanib Javed, FCPS, Principal Investigator — Ayub Teaching Hospital
Locations (1):
- Ayub teaching hospital, Abbottābād, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
will be shared after publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after publication
Access Criteria: request will be reviewed by the investigators and and further decision regarding access will be made.after publication in indexed journal it will be available online

REFERENCES:
- [Derived] Akbar I, Javed Z, Batool N. Primary versus secondary closure of stoma reversal skin wound: Randomized controlled trial. J Pak Med Assoc. 2023 Jan;73(1):4-8. doi: 10.47391/JPMA.3771. PMID 36841997